CLINICAL TRIAL: NCT04372875
Title: Leveraging Health Information Technology to Reduce Health Disparities in Adolescent Health Outcomes: A Patient-Centered Approach
Brief Title: Health Information Technology to Reduce Disparities in Adolescent Health Outcomes: A Pragmatic Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Monika Goyal, Associate Professor of Pediatrics and Emergency Medicine, Children's National Research Institute
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: Pro00014276
Record Dates: First submitted 2020-04-30; First posted 2020-05-04 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2024-12

CONDITIONS: Sexually Transmitted Diseases
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHS-derived CDS (Experimental): All adolescents seen in the emergency department that meet eligibility criteria will be offered the sexual health survey (SHS) during the pragmatic trial.
  Interventions: Behavioral: SHS-derived CDS
- Usual care (No Intervention): All adolescents seen in the emergency department that meet eligibility criteria prior to implementation of SHS-derived CDS.

INTERVENTIONS:
Behavioral: SHS-derived CDS — This intervention will provide electronic clinical decision support for adolescents who screen at risk or at high risk of an STI.
  Arms: SHS-derived CDS

SUMMARY:
We will compare differences in sexually transmitted infection (STI) detection rates between sexual health survey (SHS)-derived electronic clinical decision support (CDS) versus usual care (e.g. no provision of CDS) using an interrupted time series design. We hypothesize that population-based STI detection rates will be higher when SHS-derived electronic CDS is provided compared to usual care. Secondary analysis will include a comparison of STI detection rates by sexual risk strata (high risk vs. at risk) and race/ethnicity.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 15-21 years seeking care in the emergency department

Exclusion Criteria:

* Patients will be excluded if unable to understand English, are critically ill, cognitively impaired, or otherwise unable to provide consent for completion of the sexual health survey (SHS) and STI screening.

Ages: 15 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 18500 (Estimated)
Dates: Start 2023-03-08 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Chlamydia trachomatis (CT) / Neisseria gonorrhoeae (GC) detection rates | 3-7 days after emergency department (ED) visit
  Proportion of encounters during which patients test positive for CT/GC; measured by urine-based nucleic acid amplification tests.

SECONDARY OUTCOMES:
STI rates by race/ethnicity | 3-7 days after ED visit
  Change in STI rates by race/ethnicity

CONTACTS AND LOCATIONS:
Locations (1):
- Children's National Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No